CLINICAL TRIAL: NCT03981185
Title: Accelerated Theta Burst Stimulation for Treatment of Depression in Individuals With Detoxed Alcohol Use Disorder
Brief Title: aTBS for Treatment of Depression in AUD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled. No longer continuing with study.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gregory Sahlem, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47388
Record Dates: First submitted 2019-01-12; First posted 2019-06-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Use Disorder; Depression
Keywords: depression; TMS; transcranial magnetic stimulation; theta burst; alcohol use disorder; alcohol addiction
MeSH Terms: conditions — Alcoholism; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Accelerated theta burst treatment (Experimental): All participants will receive theta-burst TMS.
  Interventions: Device: Accelerated theta burst treatment

INTERVENTIONS:
Device: Accelerated theta burst treatment — All participants will receive iTBS (intermittent theta burst stimulation) to the left DLPFC. The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 80% of resting motor threshold adjust to the skull to cortical surface distance.
  Stimulation will be delivered to L-DLPFC using the MagPRo stimulator.

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for improvement of depressive symptoms and drinking behavior in individuals with alcohol dependence. In this open label study, all participants will receive accelerated theta-burst stimulation.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive procedure and an established technology. Research utilizing rTMS in patients with alcohol use disorder has shown some promising results. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session). Recently, researchers have aggressively pursued modifying the treatment parameters, such as using accelerated intermittent theta-burst stimulation (aiTBS), to reduce treatment times with possible enhanced efficacy with some preliminary success. This study intends to further modify the parameters to create a more rapid form of the treatment and look at the change in neuroimaging biomarkers.

ELIGIBILITY:
1. Participant aged 18-65 years old with diagnosis of alcohol use disorder.
2. Participant may also choose to or not to take pharmacotherapy during the study period.
3. Participant has tried at least one medication in the past that has not helped the alcohol use disorder. If participants are taking medication, they must be on stable psychotropic medication or psychotherapy for at least 6 weeks prior to the study with plans to continue throughout study enrollment.
4. Participant needs to be at least one week after last alcohol/ substance use and had the last drink within one year of the beginning of the study participation.
5. Participant endorses depressive symptom(s), indicated by a MARDS score >= 20.
6. All participants must be assigned to a psychiatrist and agree to continue to be assigned to a psychiatrist throughout study enrollment.
7. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline Montgomery Asberg Depression Rating Scale (MADRS) | Baseline and immediate post-stimulation
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  The MADRS uses a 0 to 6 severity scale, scored following the interview. Scoring/Interpretation: Higher scores indicate increasing depressive symptoms. ... Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.
Change from baseline Montgomery Asberg Depression Rating Scale (MADRS) | Baseline and 1 month post-stimulation
  A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  The MADRS uses a 0 to 6 severity scale, scored following the interview. Scoring/Interpretation: Higher scores indicate increasing depressive symptoms. ... Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.

SECONDARY OUTCOMES:
Change in functional connectivity from baseline as measured by MR imaging | Baseline and immediate post-stimulation
  Pre- and post resting state functional connectivity and structural T1-weighted MRI scans to determine the anti-correlated LDLPFC and SCC treatment location. The identified cluster with the greatest anti-correlation between the LDLPFC and SCC will have been utilized for the targeted aiTBS treatment. This algorithm will have also been applied to the post-imaging sessions to give measurements of voxel-wise blood flow in this anti-correlation targeted brain ROI.
Change in functional connectivity from baseline as measured by MR imaging | Baseline and 1 month post-stimulation
  Pre- and post resting state functional connectivity and structural T1-weighted MRI scans to determine the anti-correlated LDLPFC and SCC treatment location. The identified cluster with the greatest anti-correlation between the LDLPFC and SCC will have been utilized for the targeted aiTBS treatment. This algorithm will have also been applied to the post-imaging sessions to give measurements of voxel-wise blood flow in this anti-correlation targeted brain ROI.
Change in alcohol craving and consumption measured by Obsessive Compulsive Drinking Scale (OCDS) | Baseline and immediate post-stimulation
  OCDS is a 14-question self-rate tool to measure obsessive thoughts about alcohol and compulsive use of alcohol. The minimum obtainable score is 0, while the maximum obtainable score is 56. Higher scores represent a worse outcome.
Change in alcohol craving and consumption measured by Obsessive Compulsive Drinking Scale (OCDS) | Baseline and 1 month post-stimulation
  OCDS is a 14-question self-rate tool to measure obsessive thoughts about alcohol and compulsive use of alcohol. The minimum obtainable score is 0, while the maximum obtainable score is 56. Higher scores represent a worse outcome.
Change in heart rate variability | At the beginning and end of each stimulation day
  Heart rate variability will be measured using a NeuroConn device which involves electrodes being placed on the chest to record heart rate.

OTHER OUTCOMES:
Change from baseline in the Delis Kaplan Executive Function System (D-KEFS): Trail Making Test | Baseline and immediate post-stimulation
  Delis Kaplan Executive Function System (D-KEFS): Trail Making Test Description: The Trail Making Test was used to measure combined visuomotor and executive functioning including sequencing and cognitive switching. The test also provides measures of visual scanning and motor speed.
  Reference: DELIS DC, KRAMER JH, KAPLAN E, HOLDNACK J. Reliability and validity of the Delis-Kaplan Executive Function System: An update. J Int Neuropsychol Soc. 2004;10(02)
Change from baseline in the Delis Kaplan Executive Function System (D-KEFS): Trail Making Test | Baseline and 1 month post-stimulation
  Delis Kaplan Executive Function System (D-KEFS): Trail Making Test Description: The Trail Making Test was used to measure combined visuomotor and executive functioning including sequencing and cognitive switching. The test also provides measures of visual scanning and motor speed.
  Reference: DELIS DC, KRAMER JH, KAPLAN E, HOLDNACK J. Reliability and validity of the Delis-Kaplan Executive Function System: An update. J Int Neuropsychol Soc. 2004;10(02)
Change from baseline in the Hopkins Verbal Learning Test- Revised (HVLT-R) | Baseline and immediate post-stimulation
  The Hopkins Verbal Learning Test - Revised (HVLT-R) is given to assess learning and recall of verbal information. The HVLT-R is a list-learning task with three learning trials, a 20-minute delayed recall, and a recognition paradigm following the delayed recall. There are six alternate forms that allow for serial evaluation.
Change from baseline in the Hopkins Verbal Learning Test- Revised (HVLT-R) | Baseline and 1 month post-stimulation
  The Hopkins Verbal Learning Test - Revised (HVLT-R) is given to assess learning and recall of verbal information. The HVLT-R is a list-learning task with three learning trials, a 20-minute delayed recall, and a recognition paradigm following the delayed recall. There are six alternate forms that allow for serial evaluation.
Change from baseline in the Brief Visuospatial Memory Test - Revised (BVMT-R) | Baseline and immediate post-stimulation
  The Brief Visuospatial Memory Test - Revised (BVMT-R) is given to measure learning and memory of visuospatial stimuli. The BVMT-R is a task that requires the participant to learn an array of simple geometric figures over three learning trials. There is a delayed recall after 25 minutes and a recognition task following the delay. There is also a copy task following the memory recall and recognition portions of the test. There are six alternate forms that allow for serial evaluation.
Change from baseline in the Brief Visuospatial Memory Test - Revised (BVMT-R) | Baseline and 1-month post-stimulation
  The Brief Visuospatial Memory Test - Revised (BVMT-R) is given to measure learning and memory of visuospatial stimuli. The BVMT-R is a task that requires the participant to learn an array of simple geometric figures over three learning trials. There is a delayed recall after 25 minutes and a recognition task following the delay. There is also a copy task following the memory recall and recognition portions of the test. There are six alternate forms that allow for serial evaluation.
Change from baseline in the Advanced Clinical Solutions Test of Premorbid Function (TOPF) | Baseline and immediate post-stimulation
  The Advanced Clinical Solutions Test of Premorbid Function (TOPF) is given to estimate an individual's premorbid cognitive and memory functioning. Although TOPF is not impervious to the effects of cognitive dysfunction, it appears to be less affected than other measures of intellectual and memory functioning. The TOPF is based on a reading paradigm, requiring the reading and pronunciation of words that have irregular grapheme-to-phoneme translation. It does not require comprehension or knowledge of word meaning.
Change from baseline in the Advanced Clinical Solutions Test of Premorbid Function (TOPF) | Baseline and 1-month post-stimulation
  The Advanced Clinical Solutions Test of Premorbid Function (TOPF) is given to estimate an individual's premorbid cognitive and memory functioning. Although TOPF is not impervious to the effects of cognitive dysfunction, it appears to be less affected than other measures of intellectual and memory functioning. The TOPF is based on a reading paradigm, requiring the reading and pronunciation of words that have irregular grapheme-to-phoneme translation. It does not require comprehension or knowledge of word meaning.

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No